CLINICAL TRIAL: NCT00906750
Title: A Pilot Study of Flumist, a Live Attenuated Intranasal Influenza Vaccine, and Inactivated Influenza Vaccine in Children With Cancer
Brief Title: A Study of a Live Intranasal Influenza Vaccine in Children With Cancer
Acronym: FMRESP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: FMRESP
Record Dates: First submitted 2009-01-05; First posted 2009-05-21 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Cancer
Keywords: FLuMIST; Inactivated influenza vaccine; Study of FluMist versus inactivated influenza vaccine in children with cancer
MeSH Terms: conditions — Neoplasms; Influenza, Human | interventions — FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: FluMist
- 2 (Active Comparator)
  Interventions: Biological: Inactivated influenza vaccine

INTERVENTIONS:
Biological: FluMist — FluMist is a live attenuated intranasal influenza vaccine
  Arms: 1
Biological: Inactivated influenza vaccine — Inactivated influenza vaccine
  Arms: 2

SUMMARY:
Eligible research subjects will be randomized to receive either FluMist or inactivated influenza vaccine then stratified by age and necessity to receive either one or two immunizations. Subjects requiring one immunization will be immunized at Day 0. Subjects requiring two immunizations will be immunized at Day 0 and Day 28. Subjects will be observed for 30 minutes following vaccination and given a diary card to record symptoms after each vaccination.

DETAILED DESCRIPTION:
The secondary objectives of this study are to:

1. Describe the safety of FluMist and inactivated influenza vaccine.
2. Describe the incidence and duration of viral replication following immunization with FluMist.
3. To examine the association between immunization response (seroconversion or seroprotection) and baseline clinical factors (age, type of malignancy, absolute neutrophil count, absolute lymphocyte count, serum IgA, IgG and IgM levels).

ELIGIBILITY:
Inclusion Criteria:

* Age 2 through 21 (not yet reached their 22nd birthday) at the time of entry into the study
* Participant or participants parent/legal guardian available by telephone during the course of the study;
* Written informed consent (and assent, if applicable) obtained
* Currently receiving chemotherapy and /or radiotherapy for the treatment of cancer or have received chemotherapy in the past 12 weeks;
* If the participant's underlying cancer is a solid tumor, current status must be stable disease, partial response, or complete response to therapy; if the participant's underlying disease is a hematological malignancy, current status must be in remission, and if receiving chemotherapy, must be in the "continuation" or "maintenance" phase of therapy or equivalent;
* Estimated life expectancy of > 1 year

Exclusion Criteria:

* History of hypersensitivity to any component of FluMist or TIV, including egg or egg products, gelatin, or monosodium glutamate;
* History of hypersensitivity to gentamicin;
* Close contact with a severely immunocompromised patient (e.g., a hematopoietic stem cell transplant patient, during those periods in which the immunocompromised patient requires care in a protective environment
* History of Guillain-Barre´ syndrome;
* History of asthma;
* Female who is breastfeeding or lactating;

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to describe the immune response of FluMist compared with inactivated influenza vaccine in mild to moderately immunocompromised children with cancer | 6 months

SECONDARY OUTCOMES:
Immunization response | 10/31/2010
  To examine the association between immunization response (seroconversion or seroprotection) and baseline clinical factors (age, type of malignancy, absolute neutrophil count, absolute lymphocyte count, serum IgA, IgG and IgM levels).
Flumist safety | 2 years
  Describe the safety of FluMist and inactivated influenza vaccine.
Viral Replication | 1 year
  Describe the incidence and duration of viral replication following immunization with FluMist.

CONTACTS AND LOCATIONS:
Overall Officials: Silvana Carr, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Carr S, Allison KJ, Van De Velde LA, Zhang K, English EY, Iverson A, Daw NC, Howard SC, Navid F, Rodriguez-Galindo C, Yang J, Adderson EE, McCullers JA, Flynn PM. Safety and immunogenicity of live attenuated and inactivated influenza vaccines in children with cancer. J Infect Dis. 2011 Nov 15;204(10):1475-82. doi: 10.1093/infdis/jir561. Epub 2011 Sep 23. PMID 21949042
- See also: St. Jude Children's Research Hospital — http://www.stjude.org